CLINICAL TRIAL: NCT03388879
Title: Reamed Nailing Versus Taylor Spatial Frame in Tibia Shaft Fractures
Acronym: NAFTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Frede Frihagen, Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REKC 2010/1706
Record Dates: First submitted 2017-12-17; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Intervention Model Description: Prospective randomized two-group clinical trial with block randomization.
Who Masked: Outcomes Assessor
Masking Description: The researcher doing the statistical analyses will be masked for treatment Group (i.e. Group 1 or 2) in a databse blinded for treatment grioups and without variables indirectly revealing treatmnet arm. These will be analyzed later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circular frame external fixator (Experimental): A Taylor Spatial Frame should consist of 2 rings with 4 half pins/K-wire attached to each ring. If possible 3, not hydroxyapatite-coated, half pins and one K-wire should be attached to each ring. The half pins/K-wire should be spread in distance and direction for optimum stability.
  Interventions: Device: Taylor Spatial Frame
- Intramedullary nail (Active Comparator): Nailing technique according to Karladani and Styf published technique (ref: Karladani AH, Styf J. Percutaneous intramedullary nailing of tibial shaft fratures: a new approach for prevention of anterior knee pain. Injury, Int. J. Care Injury 32 (2001) 736-39)
  Interventions: Device: Intramedullary nail

INTERVENTIONS:
Device: Taylor Spatial Frame — Circular external fixator
  Other Names: Circular frame
  Arms: Circular frame external fixator
Device: Intramedullary nail — Antegrade intramedullary nail
  Arms: Intramedullary nail

SUMMARY:
This is a randomised, bi-centre, prospective, clinical trial in patients with closed tibia shaft fractures. The fracture should be fresh/acute and seen within 3 weeks after the injury. Patients will be randomised to surgery with either a Taylor Spatial Frame (Smith & Nephew, England) or a reamed intramedullar nail (according to local choice) with locking screws. Primary outcome measure is the physical component summary (PCS) of RAND Short form 36 (SF-36) after 2 years. Among secondary outcomes: Visual Analogue Scale (VAS) for pain, complications, healing, malunion, and resource use.

DETAILED DESCRIPTION:
Fractures of the lower leg (fractures of the tibia shaft with or without concurrent fracture of the fibula) are a common injury. According to our fracture register 95 patients with closed tibia fractures were operated the last 3 years at our department. Fractures with moderate or no displacement can be successfully treated with a cast and subsequent Sarmiento brace. Displaced fractures are commonly treated with an intramedullary nail. Intramedullary nailing yields a high rate of union. More than 50 % of operated patients do, however, develop chronic anterior knee pain and one third of the patients have pain at rest. This contributes a big problem for many patients both at spare time and at work. Another problem is significant rates of malunion.

The use of ring fixators utilizing rings and 1,8 mm. wires was introduced by Gavril Ilizarov more than 50 years ago, and the technique has been further developed through the introduction of six adjustable struts (Taylor Spatial Frame). This hexapod circular frame allows accurate reduction as well as a high stability. The ring fixator is less invasive and allows early weight bearing, but may be cumbersome to the patient. There is also concern about pin-tract infection, osteomyelitis and joint contracture.

Only one prior study has compared ring fixator (Ilizarov) and intramedullar nail in closed tibia fractures. The results showed significant less anterior knee pain in the patients operated with ring fixator, but the study design did not allow clear conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Closed tibia shaft fractures suited for both study treatments.
* A patient who is informed of the purpose of the investigation and who has given informed consent and willingness to accept randomisation either to Taylor Spatial Frame or intramedullary nailing.
* Willingness and ability to comply with all investigation procedures
* Age between 18 to 70 years
* Skeletally mature
* Previous unaided walking

Exclusion Criteria:

* Participation in other clinical investigations that will interfere with this study
* Mental illness or other conditions that preclude ring fixator in the judgment of the investigator
* Any other concurrent condition(s) that, in the judgment of the investigator, would prohibit the patient from participation in the study
* No other injury or previous disease that would be likely to seriously influence the long term outcome (this will exclude e.g. osteomyelitis, vascular or neurological disorder of the lower extremities, rheumatoid artist, malignancy that could influence on bone healing)
* Compartment syndrome before randomisation
* Pathologic fracture
* Ongoing or previous use the last year of drugs that can be bone anabolic (e.g. anabolic steroids, growth hormone, parathyroid hormone)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-10-31 (Actual); Primary Completion 2015-06-16 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Physical Component summary of RAND SF 36 (Short Form 36) | 24 months
  Generic Health Related Quality of Life. Mean value 50, standard deviation 10. Higher score better.

SECONDARY OUTCOMES:
Vitality Subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
Physical functioning, subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
Bodily pain, subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
General health perceptions, subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
Physical role functioning, subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
Emotional role functioning, subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
Social role functioning, subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
Mental health, subscore of RAND (SF) 36 | 6, 12, 24 months
  Generic Health Related Quality of Life. Range 0 (worst) to 100 (best).
Physical Component summary of RAND (SF) 36 | 6, 12 months
  Generic Health Related Quality of Life. Mean value 50, standard deviation 10. Higher score better.
Pain around the knee | 6, 12, 24 months
  VAS scale 0-10
Pain around the fracture site | 6, 12, 24 months
  VAS scale 0-10
Pain around the ankle | 6, 12, 24 months
  VAS scale 0-10
Complications major (composite) | 24 months
  Compartment syndrome, sequela compartment syndrome (e.g. short foot, clawing, neurological disorder), infection that needs operation, any unexpected reoperation (except removal of single pins or screws)
Complications minor (composite) | 24 months
  pin tract infection that needs antibiotics, wound complication that don't need reoperation, unexpected minor reoperations (i.e. removal of single pins or screws)
Reoperations minor (composite) | 6, 12, 24 months
  Minor reoperation (e.g. remove/exchange pins, remove/exchange screws)
Reoperations major (composite) | 6, 12, 24 months
  Major reoperation (e.g. fasciotomy, exchange nail, surgery for refracture, revision for infection, surgery for non-union)
Time to union (composite) | 6, 12, 24 months
  Time to fracture union in days. We require both radiographical union defined by callus bridging 3 of 4 cortices AND clinical union defined by full, pain free and unaided weight bearing.
Resource use; Away from work | 24 months
  Number of days away from work for employed patients
Resource use; Emergency contacts | 24 months
  Number of unscheduled contacts with hospital regarding tibia fracture
Resource use; Length of stay | 24 months
  Hospital stay in days for index stay
Resource use; Operation time | 24 months
  Surgery time in minutes for index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jan E Madsen, PhD, Study Chair — Professor, head of research group
Locations (1):
- Orthopedic Center, Ulleval University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Depending on demand. No plan as of yet.